CLINICAL TRIAL: NCT07327658
Title: Investigation of the Changes in Periodontal Pocket Depth Following Periodontal Treatment in Patients With Periodontitis
Brief Title: Changes in Periodontal Pocket Depth After Periodontal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Osman Babayigit, Asistant Professor, Necmettin Erbakan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-DIS-OB-04
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis
Keywords: Periodontitis; Periodontal Therapy; Periodontal Pocket
MeSH Terms: conditions — Periodontitis; Periodontal Pocket | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-Surgical Periodontal Treatment (Experimental): Participants with periodontitis received non-surgical periodontal treatment. Periodontal pocket depth was recorded at baseline and at 1, 3, and 6 months following treatment.
  Interventions: Procedure: Periodontal Treatment

INTERVENTIONS:
Procedure: Periodontal Treatment — Periodontal treatment was performed according to standard clinical protocols. Periodontal pocket depth was measured at baseline and at 1, 3, and 6 months following treatment.

SUMMARY:
This study is a prospective, observational clinical research conducted at the Department of Periodontology, Faculty of Dentistry, Necmettin Erbakan University. The study aims to evaluate periodontal records routinely obtained before treatment and throughout the treatment process from individuals who visited the clinic and were planned for non-surgical periodontal treatment. Within the scope of the research, the effectiveness of periodontal treatments will be evaluated solely through non-invasive clinical periodontal parameters. No additional invasive procedures will be performed during the study; only records obtained during routine periodontal examinations and treatments at the clinic will be used.

DETAILED DESCRIPTION:
Patient Selection:

The study will include individuals aged 18-65 who have been diagnosed with periodontitis. All patients' treatment processes will be carried out within the framework of standard protocols implemented at our clinic, and patients will be called for regular follow-up appointments scheduled between 1 month and 1 year after treatment. Data from patients with a 6-month follow-up period will be evaluated within the scope of the study.

Inclusion Criteria:

* Aged 18-65
* Not pregnant or breastfeeding
* Smoking less than 10 cigarettes per day
* Diagnosis of periodontitis in clinical records (stage 3 and 4 according to the 2017 classification)

Exclusion Criteria:

* Individuals with uncontrolled systemic disease
* Patients diagnosed with diabetes
* Individuals under 18 years of age
* Individuals who smoke 10 or more cigarettes per day
* Patients who do not attend regular follow-up appointments and do not have sufficient clinical records

Clinical Periodontal Examination and Measurements:

All individuals participating in the study undergo routine clinical and radiographic evaluations before and during treatment. The parameters measured during periodontal examinations are as follows:

* Periodontal pocket depths
* Clinical attachment levels
* Bleeding index on probing
* Gingival index
* Plaque index
* Keratinized gingival width
* Tooth mobility and furcation defect grades
* Gingival recession

Patients' sociodemographic data and oral hygiene habits are also recorded. Periodontal disease diagnosis and classification are performed according to the 2017 Classification of Periodontal and Peri-Implant Diseases and Conditions criteria.

Stage 3 periodontitis: 25 individuals Stage 4 periodontitis: 25 individuals

Application Principle of the Study:

No additional interventional procedures will be performed on individuals within the scope of this study; records obtained during routine treatments at the clinic will be used. The effectiveness of periodontal treatments will be evaluated by comparing clinical measurements obtained before periodontal treatment and during follow-up sessions. The main objective of the study is to demonstrate the effectiveness of non-surgical periodontal treatment protocols through the analysis of clinical records.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age
* Not being pregnant or breastfeeding
* Smoking less than 10 cigarettes a day
* Having a clinical record of periodontitis (stages 3 and 4 according to the 2017 classification)

Exclusion Criteria:

* Individuals with uncontrolled systemic disease
* Patients diagnosed with diabetes
* Individuals under 18 years of age
* Individuals who smoke 10 or more cigarettes a day
* Patients who do not attend regular follow-up appointments and do not have sufficient clinical records

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Change in Periodontal Pocket Depth | Baseline, 1 month, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology, Konya, Turkey, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Citterio F, Kanmaz B, Baima G, Romano F, Buduneli N, Aimetti M. Pocket closure in stage III-IV grade C periodontitis: A multilevel analysis following non-surgical periodontal therapy. Int J Dent Hyg. 2024 Aug;22(3):547-553. doi: 10.1111/idh.12688. Epub 2023 May 8. PMID 37154234